CLINICAL TRIAL: NCT02579044
Title: Phase I/II Trial of Everolimus in Combination With Lonafarnib in Progeria
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Monica E. Kleinman, Medical Director, Transport & MSICU, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00017505
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Progeria
MeSH Terms: conditions — Progeria | interventions — Everolimus; lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus and Lonafarnib (Other): Single arm. Phase I: Lonafarnib with escalating doses of everolimus to determine MTD Phase II: Lonafarnib plus everolimus at MTD (efficacy assessment)
  Interventions: Drug: Everolimus and lonafarnib

INTERVENTIONS:
Drug: Everolimus and lonafarnib

SUMMARY:
This is a phase I/II dose-escalation trial of everolimus in combination with lonafarnib in Hutchinson-Gilford Progeria Syndrome (HGPS) and progeroid laminopathies (henceforth "progeria"). The study will be conducted at a single clinical site utilizing the Clinical and Translational Study Unit (CTSU) at Boston Children's Hospital. Lonafarnib will be administered at doses previously established in the pediatric population and in this population of progeria subjects. This study will first determine the dose-limiting toxicities (DLT) and the maximum tolerated dose (MTD) of everolimus when administered in combination with lonafarnib. It will then determine the efficacy of everolimus when administered at its MTD in combination with lonafarnib for disease in progeria.

ELIGIBILITY:
Inclusion Criteria:

* Genetically-confirmed progeria.
* display clinical signs of progeria as per the clinical trial team.
* currently receiving lonafarnib under protocol 09-06-0298
* have not experienced a grade 3 or 4 toxicity within two months preceding enrollment
* willing and able to come to Boston for appropriate studies and examinations.
* no recent fractures or major surgery (within four weeks)
* Absolute poly count (Absolute neutrophil count + bands + monocytes) >1,000/uL
* platelets >75,000/uL (transfusion independent)
* hemoglobin >9 g/dL
* creatinine ≤ 1.5 times upper limit of normal (ULN) for age or Glomerular filtration rate (GFR) >70 mL/min/1.73m2
* bilirubin ≤ 1.5x upper limit of normal for age
* SGPT (ALT) < and SGOT (AST) ≤ 2.5x normal range for age
* serum albumin greater than or equal to 2 g/dL
* PT/PTT: INR <1.3 (or <3 on anticoagulants)
* Fasting LDL cholesterol within 1.5x ULN per institutional guidelines (ie, <195 mg/dL for 2 - 18 years of age, <240 mg/dL for subjects >18 years old)* and Fasting serum cholesterol <300 mg/dL (<7.75 mmol/L)* and Fasting triglycerides <2.5 ULN (<325 mg/dL for ages 2 - 18, <400 for ages >18)*

  *may be re-evaluated for eligibility after initiation of lipid-lowering therapy
* Signed informed consent according to institutional guidelines must be obtained and subject must begin therapy within twenty-eight (28) days.

Exclusion Criteria:

* Subjects must not be taking medications that significantly affect the metabolism of lonafarnib
* Subjects receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Subjects with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary. Topical or inhaled steroids are allowed.
* Subjects who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug; have not recovered from the side effects of any major surgery (defined as requiring general anesthesia but excluding a procedure for insertion of central venous access); or who may require major surgery during the course of the study.
* 13.2.5 Subjects with an active bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin).
* Subjects who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * known severely impaired lung function
  * active (acute or chronic) or uncontrolled severe infections.
  * liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
  * History of hepatitis B or hepatitis C
* Other concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration).
* A known history of Human Immunodeficiency Virus (HIV) seropositivity or known immunodeficiency.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A nasogastric tube (NG tube) or gastric tube (G tube) is allowed.
* Subjects who have known or suspected hypersensitivity to any of the excipients included in the formulation should not be treated.
* Subjects must not be pregnant or breast-feeding. Female subjects of childbearing potential must have negative serum or urine pregnancy test. Sexually active male and female subjects of reproductive potential must agree to use a medically accepted form of birth control while on study and up to 10 weeks after treatment. It is permissible for female subjects to take oral contraceptives or other hormonal methods while receiving treatment with everolimus.

Ages: 18 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of everolimus when administered orally in combination with lonafarnib in subjects with progeria | 12 Months
  For Phase I portion of protocol
Number and type of dose-limiting toxicities when everolimus and lonafarnib are administered in combination to children with progeria | 12 Months
  For Phase I portion of protocol
Annual increase in weight gain | 24 Months
  For Phase II portion of protocol
Change in pulse wave velocity (PWV) | 24 months
  For Phase II portion of protocol

SECONDARY OUTCOMES:
Markers of progeria-specific activity | 24 Months
  For Phase II portion of protocol
Trough levels of everolimus in combination with lonafarnib in progeria | 12 months
  For Phase I portion of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Monica Kleinman, M.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States